CLINICAL TRIAL: NCT01824511
Title: Does Smoking Cessation Increase Anhedonia? A Test of Pre-clinical Findings
Brief Title: Effects of Quitting Study A Test of Pre-clinical Findings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Hughes, Principal Investigator, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHRBS B11-185; R01DA031687 (NIH)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Smoking
Keywords: smoking; nicotine; tobacco; anhedonia; reward; withdrawal
MeSH Terms: conditions — Smoking; Anhedonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smokers Cease Smoking (Experimental): Participants are paid to quit smoking without using any medications.
  Interventions: Behavioral: Smokers cease smoking

INTERVENTIONS:
Behavioral: Smokers cease smoking — Smokers are paid to be abstinent for four weeks, and stop-smoking medications may not be used.

SUMMARY:
The most widely-accepted animal model of nicotine withdrawal states stopping nicotine makes rewarding events become less rewarding. The current study will test if this is true in humans. If we find tobacco abstinence does make rewards less rewarding, this would suggest new symptoms to add to official descriptions of nicotine withdrawal. It would also suggest we need to develop new behavioral and pharmacological interventions to correct this problem. If stopping smoking does not make rewards less rewarding, this would suggest this animal model does not apply to the human condition and we need to continue to search for an animal model of tobacco withdrawal that is relevant to smokers stopping smoking.

DETAILED DESCRIPTION:
Study design We will recruit until we have 70 current smokers who want to quit at two sites (Univ of Vermont and Dartmouth Medical School). We will also recruit a comparison group of 70 long-time former smokers to assist in interpretation of the results. In the first week, smokers will smoke their usual number of cigs/day. They will then quit and are to remain abstinent for 4 weeks. We will use a schedule of escalating monetary contingencies based on breath and saliva and/or urine samples to encourage abstinence. We will obtain dependent measures twice/week. The primary measures of reward responsivity will be the percent choosing the hard task and the amount of responding for a monetary reward on the EEfRT task and the score on our Rewarding Events scale. Other outcomes will be delay discounting results and self-reports of anhedonia and apathy.

The study will run for 1 week pre-cessation (2 visits) and then for 4 weeks post-cessation. Measures and biochemical verifications will occur twice/wk. Former smokers will attend once a wee for four weeks.

For the first week of abstinence, the cutoff for nonsmoking will be CO <8 ppm. For the remaining weeks, abstinence will be verified with a score of 0 (<10 ng/ml of cotinine) on a test strip in a saliva or urine sample plus a CO <8 ppm.

At the initial session, completion of baseline surveys will describe the sample and also measure plausible moderators such as depression.

We believe the most direct test of reward sensitivity is an evaluation of the influence of abstinence on operant responding for a reward. Thus, we have chosen performance on the Effort Expenditure for Rewards Task (EEfRT), which examines responding as a function of response cost, reward magnitude and probability of reward, as one of our primary outcomes.

For a self-report measure we will use our Rewarding Events (RE) scale that asks both about occurrence of presumed rewarding events and their anticipated pleasantness. Our RE scale will ask participants to rate 58 items on frequency in the last week as well perceived/expected pleasantness of events.

Secondary measures include the 18-item Apathy Evaluation Scale (AES), the Temporal Experience of Pleasure (TEPS), Minnesota Nicotine Withdrawal Scale-Revised (MNWS), and a measure of delay discounting (DD).

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* 18 yrs old or older
* able to read and understand verbal English fluently
* citizen or resident alien
* agree to abstain from illegal drugs during the study

For current smokers:

1. currently smoke >10 cigarettes daily for > 1 yr
2. want to quit smoking for good via abrupt cessation without treatment
3. willing to quit 7-14 days from study entry and not reduce before quitting
4. no reduction in cigs/day by >25% in the last month
5. agree to no use of non-cigarette tobacco, non-tobacco nicotine, marijuana, illegal drugs, electronic cigarettes, or smoking cessation medications during the study
6. have carbon monoxide (CO) level > or = 8 ppm at the time of consent
7. no current use of prescribed psychoactive medications, including smoking cessation products.

For former smokers:

1. smoked >10 cigarettes daily for > 1 yr
2. quit at least 1 yr ago
3. use of cigarettes or e-cigarettes 5 or fewer times in past year
4. no tobacco or nicotine-containing product in last month
5. agree to no use of non-cigarette tobacco, non-tobacco nicotine, marijuana, illegal drugs, electronic cigarettes, or smoking cessation medications during the study
6. have carbon monoxide (CO) level < 8 ppm at the time of consent
7. no current use of prescribed psychoactive medications, including smoking cessation products.

Exclusion Criteria for all participants:

* History of hand or wrist problems that could be exacerbated by study participation or interferes with completion of tasks
* current (last year) mood or alcohol/drug-related psychiatric disorder or any neurological condition that could influence reward sensitivity; e.g. Parkinsonism
* used marijuana 2 or more times in the last month
* problems with the use of alcohol or illegal drugs in the last 6 months
* currently pregnant
* use of smokeless tobacco
* lacking the use of one or both hands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Responses to Effort Expenditure for Rewards Task (EEfRT) Test | four weeks after quit date
  The primary outcome will be the percent choosing the hard task and the amount of responding for a monetary reward on the EEfRT task.
Rewarding Events Scale score. | four weeks after quit date
  The score on our Rewarding Events scale.

SECONDARY OUTCOMES:
Delayed Discounting | four weeks after quit date
  Measures preference for immediate vs. delayed rewards by responses to several scenarios. Outcome is a statistic that describes relative preference by time to reward.
Self-reports of Anhedonia and Apathy | four weeks after quit date
  Temporal Experience of Pleasure (TEPS) and Apathy Evaluation Scale (AES) both ask participants to rate pleasantness of common rewards. Outcome is mean rating on ordinal scales. Positive and Negative Affect Scale (PANAS) and the Minnesota Nicotine Withdrawal Scale-Revised (MNWS) ask participants to rate several mood or nicotine withdrawal symptoms. Outcome is mean rating on 4 or 5 point ordinal scale.

CONTACTS AND LOCATIONS:
Overall Officials: John R Hughes, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Dartmouth College, Hanover, New Hampshire
  - University of Vermont, Burlington, Vermont